

Version Date: September 2, 2023

TO: ALL NATIONAL CLINICAL TRIALS NETWORK (NCTN) MEMBERS AND NCI

COMMUNITY ONCOLOGY RESEARCH PROGRAM (NCORP) AFFILIATES AND

SUBAFFILIATES; CTSU

FROM: SWOG Operations Office (<u>protocols@swog.org</u>)

RE: <u>\$1826</u> "A Phase III, Randomized Study of Nivolumab (Opdivo) Plus AVD or

Brentuximab Vedotin (Adcetris) Plus AVD in Patients (Age >/= 12 Years) with Newly Diagnosed Advanced Stage Classical Hodgkin Lymphoma" Study Chairs: Drs. A. F. Herrera, J. Friedberg, S. M. Castellino, S. Parsons, S. C. Rutherford, A. M. Evens, A. Punnett, K. Davison, D. Hodgson, L. S. Constine, L. Kostakoglu Shields, J. Y. Song.

#### **REVISION #6**

Study Chair: Alex F. Herrera, M.D. Phone number: 626/256-4673 E-mail: <a href="mailto:aherrera@coh.org">aherrera@coh.org</a>

#### **Action Codes**

 $(\sqrt{})$  Expedited review allowed

#### **Key Updates**

(√) Eligibility changes\*

\*Patient notification not required

 $(\sqrt{})$  Data Submission changes

 $(\sqrt{})$  Editorial / Administrative changes

**Sites using the CIRB as their IRB of record**: The protocol and/or informed consent form changes have been approved by the CIRB and must be activated within 30 days of distribution of this notice through the CTSU Bi-Monthly Broadcast email.

Sites not using the NCI CIRB: Per CTMB Guidelines, the protocol updates and/or informed consent changes must be approved by local IRBs within 90 days of distribution of this notice through the CTSU Bi-Monthly Broadcast email. The changes are effective upon approval by the local IRB; however, any changes to eligibility are effective 30 days after distribution of this notice. If local IRB approval is not granted within 30 days, new registrations must meet any revised eligibility criteria included in the revision or accrual must be suspended until approval is obtained.

#### **REVISION #6**

The above referenced study has been revised to: (1) primarily ask sites to submit two additional, previously collected, scans based on protocol specifications; (2) Expand eligibility. The changes are as follows:

#### **Protocol Changes**

- 1. The version date has been updated.
- Throughout the protocol, formatting, typographical errors, pagination, and cross-references have been corrected as needed.

- 3. <u>Section 5.6a:</u> This section has been expanded upon to include, "Patients who do not complete PRO instruments prior to registration but are otherwise eligible will remain eligible for the primary analysis and other secondary analyses" to maintain eligibility for patients.
- 4. **Section 9.2:** Footnote "e" was edited to emphasize CT scan requirements.
- 5. **Section 13.5g:** The request for Patient SSN information was removed.
- 6. <u>Section 14.4a:</u> The location of the Imaging Adjunctive Data Sheet link was updated.
- 7. <u>Section14.4f:</u> This section has been inserted to include, "All contrast-enhanced CT images involved at baseline or contraindicated from scans performed to assess disease as specified in Section 15.4. Submit to IROC Ohio (via TRIAD strongly preferred) for retrospective central imaging review."
  - The location of the Imaging Adjunctive Data Sheet links were updated.
  - For patients who have had 1-year and 2-year after registration contrast-enhanced CT (or if contra-indicated, PET-CT, CT, MRI, or MR-PET) scan performed prior to activation of S1826 Protocol Revision 6, submit images to IROC Ohio within 60 days after participating site activation of S1826 Protocol Revision 6 (Version Date 9/2/2023).
  - If CT scan is contraindicated and PET-CT scan is submitted, S1826 Imaging Adjunctive Data Sheet for PET scans is required. This form is submitted electronically via the IROC website.
- 8. **Section 15.4a:** Under Image Collection and Submission Time Points:
  - "If performed" was removed from criterion 4.
  - Criteria 5 and 6 were inserted to indicate the required scan submissions as 1 and 2 years after registration, respectively.

#### **Consent Changes**

- 1. The version date has been updated.
- 2. Throughout the consent, formatting, typographical errors, pagination, and cross-references have been corrected as needed.
- 3. The reading scores were updated.
- 4. <u>"What exams, tests, and procedures are...":</u> Under the subheader, "For both Groups 1 and 2,":
  - In the seventh bullet regarding Patient Reported Outcomes, language requiring patient reported outcomes for participation in the overall study was removed.
  - o In the eighth bullet regarding patient scans, patients are informed that scans from their 1<sup>st</sup> and 2<sup>nd</sup> years after registration will be submitted to the study for review.

#### Patient Notification and use of Consent Addendum:

Please note that the information provided below regarding patient notification and amendments to local consent forms reflects SWOG's minimum requirements. Sites should refer to the policies/procedures of the IRB of record to determine whether they have any more stringent requirements.

SWOG has determined that the changes above that are **bolded** may affect a patient's willingness to participate in the study; therefore, SWOG requires that patients be notified of these changes.

Who must be informed?

• All patients who have been consented to the study and received treatment.

How must patients be notified?

• Notification must take place either via the attached Consent Addendum or via amended consent form by next study visit. After the change has been discussed with the patient, the patient must sign and date either the Consent Addendum or the [Publish Date] version of the consent form.

What is the notification deadline and process?

- Patients must be notified by their next scheduled visit or within 90 days after CTSU distribution of this revision, whichever is sooner.
- <u>Sites using the NCI CIRB as their IRB of record</u>: CIRB has approved the attached Consent Addendum; therefore, the Consent Addendum may be utilized immediately to notify patients of these changes.
- Sites not using the NCI CIRB as their IRB of record: If local IRB approval of the Consent Addendum is required before sites may utilize it, the site must still notify patients verbally prior to the notification deadline and notification must be documented in the patient chart. The site must then obtain patient signature on the Consent Addendum or updated consent form once the addendum and/or revised consent is locally approved. Important: Any changes to eligibility criterion are effective 30 days after distribution of this notice. If local IRB approval is not granted within 30 days, new registrations must meet any revised eligibility criteria included in the revision or accrual must be suspended until approval is obtained.

#### Regulatory Considerations:

Do local consent forms need to be updated?

• Yes, local consent forms must be updated to include all the changes in this revision.

The updated protocol and model informed consent form can be accessed from the CTSU website (<a href="www.ctsu.org">www.ctsu.org</a>). Please discard any previous versions of the documents and replace with the updated versions. Please contact lymphomaquestion@crab.org or 206/652-2267 with any questions.

This memorandum serves to notify the NCI, and SWOG Statistics and Data Management Center.

PROTOCOL & INFORMATION OFFICE CC: Hildy Dillon, MPH - Patient Advocate Sharon M. Castellino, MD, MSc - COG Susan K. Parsons, MD, MRP - COG Angela Punnett, MD, FRCPC - COG Catherine Shannon - COG Tiffany Liu, MS, MA - COG Sarah C. Rutherford, MD - Alliance Andrew M. Evens, MD - ECOG-ACRIN Kelly Davison, MD - CCTG Michael Crump, MD - CCTG Joo Y. Song, MD - Pathology Louis S. Constine, MD, FASTRO, FACR - Radiation Oncology David Hodgson, MD - Radiation Oncology Lale Kostakoglu Shields, MD, MPH - Radiology

# **Informed Consent Addendum Model for <u>\$1826</u>**

S1826, "A Phase III, Randomized Study of Nivolumab (Opdivo)
Plus AVD or Brentuximab Vedotin (Adcetris) Plus AVD in Patients
(Age >/= 12 Years) with Newly Diagnosed Advanced Stage Classical
Hodgkin Lymphoma"

The following information should be read as an update to the original Consent form that you read and signed at the beginning of the study. Unless specifically stated below, all information contained in that original Consent Form is still true and remains in effect. Your participation continues to be voluntary. You may refuse to participate, or may withdraw your consent to participate at any time, and for any reason, without jeopardizing your future care at this institution or your relationship with your study doctor.

## New or additional information

The consent form has been updated to include two additional scan reports you've already had as part of your care. We are requesting the two new reports from one and two years after you joined the study. There will be no extra appointments as these scans are already done.

## **Patient Signature and Date**

By signing this form, I acknowledge that I have read the information above or had it read to me. I have discussed it with a member of the study team and my questions have been answered. I understand that I will be given a copy of this form.

| Participant's signature |
|-------------------------------------------------------------------|
| Date of signature |
| Signature of person(s) conducting the informed consent discussion |
| Date of signature |

Readability Statistics:

Flesch Reading Ease: 61.4 (targeted above 55)

Page 1

Flesch-Kincaid Garde Level 9.2 (targeted below 8.5)

Version Date 9/2/2023

# **Research Study Informed Consent Document**

Study Title for Study Participants: Testing nivolumab plus the standard chemotherapy in comparison to brentuximab vedotin plus the standard chemotherapy for Newly Diagnosed Advanced Stage Classical Hodgkin Lymphoma

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:
A Phase III, Randomized Study of Nivolumab (Opdivo) Plus AVD or
Brentuximab Vedotin (Adcetris) Plus AVD in Patients (Age >/= 12 Years)
with Newly Diagnosed Advanced Stage Classical Hodgkin Lymphoma

If you are a parent or legal guardian of a child who may take part in this study, permission from you is required. The assent (agreement) of your child may also be required. When we say "you" in this consent form, we mean you or your child; "we" means the doctors and other staff.

# **Overview and Key Information**

# What am I being asked to do?

We are asking you to take part in a research study (clinical trial). This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this study because you have been recently diagnosed with advanced stage classical Hodgkin Lymphoma.

# Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

This study is being done to answer the following question: If we add the study drug nivolumab to standard chemotherapy will it extend your time without disease more than or less than if we add the study drug brentuximab vedotin to standard chemotherapy? We will also compare any side effects you may have and your well-being when you take the study drugs and for up to ten years after you stop taking these drugs to treat the cancer.

## What is the usual approach to treat classical Hodgkin Lymphoma?

These treatments have been approved by the Food and Drug Administration (FDA). The usual approach for children and adolescents who are not in a study is treatment with standard chemotherapy, which may be followed by radiation therapy. Chemotherapy is a name for drugs that fight cancer cells. Radiation therapy is the use of high energy x-rays to kill cancer cells. There are several chemotherapy drugs approved by the FDA that are commonly used with the radiation therapy. For patients who receive the usual approach for this cancer, about 70-80 out of every 100 patients are free of cancer at five years.

# What are my other choices if I do not take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.

# What will happen if I decide to take part in this study?

Adults, children and adolescents who are part of this study will be treated in 1 of 2 ways. You will get either nivolumab plus the usual three chemotherapy drugs (doxorubicin, vinblastine, and dacarbazine, which is also known as AVD), or brentuximab vedotin plus the usual three chemotherapy drugs (AVD). You will also have tests during your treatment to see if the cancer is getting worse, staying the same, or getting better. Depending upon how the cancer responds to the study drugs, you may also receive radiation therapy as part of your treatment.

If you decide to take part in this study, you will get either the study drug nivolumab plus standard chemotherapy for up to 6 cycles, or you will get the study drug brentuximab vedotin plus standard chemotherapy for up to 6 cycles. After you finish the chemotherapy cycles, your treating physician may decide to give you radiation therapy based on the tumor response at time of completion of all 6 cycles of chemotherapy.

After you finish your treatment (chemotherapy and, for some people, radiation therapy), your doctor and study team will watch you for side effects. They will check you every 3 months for the first year from the time you began this study. After that, they will check you every 6 months for the second and third years after you began this study, and then they will check you once a year for the fourth through tenth years. This means you will keep seeing your doctor for 10 years after you begin treatment.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the addition of the study drugs may not be as good as the usual approach for the cancer.

There is also a risk that you could have side effects from the study drugs. These side effects may be worse and may be different than you would get with the usual approach for the cancer.

Some of the most common side effects from the study drugs that doctors know about are:

- Low blood pressure which may cause dizziness or high blood pressure which may cause headaches, dizziness or blurred vision
- Anemia, which may require transfusion
- Tiredness or difficulty sleeping
- Bruising or bleeding
- Nausea, vomiting, diarrhea, constipation, loss of appetite
- Infection, especially when white blood cell count is low, chills, fever, body aches or Muscle Pain
- Pain, pain in belly, pain or swelling of the joints, or pain or redness at the site of injection
- Numbness, tingling or pain of the arms and legs
- Mouth sores or dry mouth
- Muscle weakness

There may be some risks that the study doctors do not yet know about. More information about risks will be provided below (beginning on Page 7).

#### **Benefits**

There is evidence that the study drugs are effective in shrinking your type of cancer. This study will help the study doctors learn things that will help people in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

# Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women of childbearing potential: You become pregnant while on the study.
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (SWOG Cancer Research Network). The study sponsor is the organization that oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

# What is the purpose of this study?

The purpose of this study is to compare nivolumab plus the three chemotherapy drugs: doxorubicin, dacarbazine, and vinblastine sulfate (AVD) to brentuximab vedotin plus the three chemotherapy drugs: doxorubicin, dacarbazine, and vinblastine sulfate (AVD), followed by targeted radiation therapy in some patients with lymphoma that does not completely respond to therapy. The addition of either nivolumab or brentuximab vedotin to the usual treatment could shrink the cancer or extend your time without your disease symptoms coming back. But, it could also cause side effects, which are described in the risks section below.

Nivolumab is an immunotherapy drug (a type of drug that works by boosting your immune system) that attaches to a target protein called PD-1 (found within white blood cells) and helps to increase the immune system's activity against the cancer. Brentuximab vedotin is an antibody drug conjugate, which means that the drug contains an antibody that attaches to a protein (CD30) that is found on the surface of classical Hodgkin Lymphoma cells and then releases a drug inside those cells that kills the cancer cells.

This study will help the study doctors find out if one of the drug combinations (nivolumab plus the usual chemotherapy or brentuximab vedotin plus the usual chemotherapy) is better, the same, or worse than the other drug combination, followed by radiation therapy in some patients. To decide if it is better, the study doctors will be comparing the drug combinations to see which drug combination allows more patients to have no disease symptoms at 2 years or more after the completion of the study treatment and which drug combination extends the overall survival of patients at 10 years after completion of the study treatment.

Nivolumab is already approved by the Food and Drug Administration (FDA) for the treatment of relapse or progression of classical Hodgkin lymphoma after stem cell transplant and treatment with either brentuximab vedotin or 3 lines of systemic therapy. Nivolumab is not approved by the FDA for use in newly diagnosed patients (of any age) with classical Hodgkin lymphoma.

Brentuximab vedotin is approved by the FDA for the treatment of newly diagnosed advanced classical Hodgkin lymphoma, when added to chemotherapy (including AVD), in adult patients. Brentuximab vedotin is not approved by the FDA for the same use in patients under 18 years of age.

There will be about 987 people taking part in this study.

# What are the study groups?

This study has two study groups.

# Group 1

Group 1 will receive nivolumab plus three chemotherapy drugs (doxorubicin, vinblastine, and dacarbazine) by intravenous infusion on Day 1 and Day 15 of each cycle (every 2 weeks for a total of 6 cycles). A cycle is every 28 days. You will not have to be in the hospital for the drug infusion unless your doctor feels it is needed. Your doctors may also recommend radiation therapy at the end of 6 cycles of treatment.

#### Group 2

Group 2 will receive brentuximab vedotin plus three chemotherapy drugs (doxorubicin, vinblastine, and dacarbazine) by intravenous infusion on Day 1 and Day 15 of each cycle (every 2 weeks for a total of 6 cycles). A cycle is every 28 days. Your doctors may also recommend radiation therapy at the end of 6 cycles.

## Both Groups 1 and 2:

Filgrastim and pegfilgrastim are drugs that are used to prevent the white blood cell count from dropping too low after treatment in order to avoid infections. If you are in Group 2, you will receive either filgrastim or pegfilgrastim (as indicated below) to prevent infection as part of the study treatment. If you are in Group 1, you may receive filgrastim or pegfilgrastim (as indicated below) if your physician recommends it to prevent infection.

- If you receive pegfilgrastim, it will be given on Day 2 and Day 16 via an injection under the skin. Your doctor may give you an injector kit to wear to receive this drug.
- If you are an adult and you receive filgrastim, it will be given for about 2-5 days (such as, on Days 6-10 and Days 21-25) via an injection under the skin or via intravenous (IV) infusion.
- If you are younger than 18 years of age and you receive filgrastim (via an injection under the skin or via intravenous (IV) infusion), it will be given every day, beginning on Day 4, 5, 6, 7, 8, or 9 and will continue for as many days as recommended by your doctor. If you are still receiving filgrastim on Day 14, it will be stopped on Day 14 (24 hours prior to your receiving the study drugs on Day 15) and it may be started again Day 16.

You will receive study drug for up to approximately 6 months. After you complete all 6 cycles of chemotherapy, if your study doctor recommends radiation therapy, then you may also receive radiation therapy for approximately 1 month.

We will use a computer to assign you to one of the study groups. This process is called "randomization." It means that your doctor will not choose and you cannot choose which study group you are in. You will be put into a group by chance. You will have an equal chance of being in Group 1 or Group 2.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.



You will be asked to fill out up to 3 questionnaires at 5 timepoints:

prior to beginning the study, on Day 1 of Cycle 3,

within 4-8 weeks after completion of treatment,

1 year after you begin the study and 3 years after you begin the study.

You will also be asked to fill out 1 questionnaire at up to 14 timepoints.

# What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health that may not be included in the usual care (if you were not in this study). We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects. These extra exams, tests, and procedures to monitor your safety and health include:

To take part in this study there must be available tissue left over from a biopsy done at the time of cancer diagnosis to submit to the study for central review by the study doctors. PET/CT scans are a way to take pictures of classical Hodgkin Lymphoma. Your doctor will be required to submit images of your PET/CT scans (that are done at 2-3 timepoints for the usual care for your cancer) for review by the study doctors. The results of these reviews will not be shared with you or your doctor.

## For Group 1 only:

• You will have a blood test on Day 1 of every other cycle to check your thyroid function.

#### For both Groups 1 and 2:

- If you are a woman who can have children, a pregnancy test before you start the study.
- If you are HIV-positive, a blood test to check your HIV viral load and CD4 count (to ensure it is safe for you to receive study drugs) before you start the study.
- Blood tests done on Day 1 and Day 15 of each cycle of treatment to check your health and organ function.
- Physical exams done on Day 1 of each cycle of treatment.
- Your study doctor will need to use some of the tissue left over from your biopsy when you were diagnosed with cancer. This sample is a required part of the study. There must be tissue available from the biopsy done at time of your diagnosis to take part in this study. The doctor that ordered the biopsy will send a tissue slide or block to the study doctors, so that the study doctors can confirm that they agree with your diagnosis. Because this review by the study doctors is done later (and possibly after completion of your study treatment), you and your study doctor will not get the results of this testing.
- In addition to the slides submitted to the central lab for testing, you will asked to agree or not agree to have a tissue block or slides submitted for banking for future studies. You can indicate whether you will allow your specimens to be banked for future studies in the section called "Optional Studies".
- You will be asked to fill out up to 3 forms at 5 timepoints (prior to beginning the study, Day 1 of Cycle 3, within 4-8 weeks after your last dose of study drug, 1 year after you start the study and 3 years after you start the study). You will also be asked to fill out 1 form at up to 14 timepoints (Day 1 of each cycle, within 4-8 weeks after your last dose of study drug, 3-6 month follow-up visit after you start the study (if you go off treatment early), and 9, 12, 18, 24, 30, and 36 months after you start the study. All of the forms will take a total of about 30 minutes to complete. The forms will ask questions about your health (physical and emotional well-being), any side effects that you may have related to the cancer treatment and your well-being. You don't have to answer any question that makes you feel uncomfortable. Researchers will use this information to learn more about classical Hodgkin Lymphoma and how the treatments in this study affect people.

Important: Since these forms are being used for research, the responses you provide will not be shared with your study doctor. If you have any serious health issues or other concerns, please talk with your doctor or nurse right away.

• As part of your usual care, your doctors look at PET/CT scans, which are a way to take pictures of your type of cancer. For both Groups 1 and 2, your doctor will be required to submit copies of your PET/CT scans for review by the study doctors. Scans will be submitted: before you started the study drugs, at the end of Cycle 2 (if your doctor ordered a scan), and within 4-8 weeks after you complete all 6 cycles of the study drugs. If you received a scan at 1 and 2 years after registration, these will also be submitted for review by the study doctors.

# What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the study drugs may not be as good as the usual approach for your cancer at preventing the cancer from progressing or from coming back after treatment.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The study drugs (and possible radiation therapy) used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and after you complete the study treatment. For women: Do not get pregnant or breastfeed while taking part in this study or for 6 months after you receive the last dose of study drug or after your last dose of radiation therapy (if applicable). For men: Do not father a baby while taking part in this study or for 7 months after you receive the last dose of study drug or for 6 months after your last dose of radiation therapy (if applicable). For all: Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 7 months after your last dose of study drug.

This study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat this type of cancer in the future. Because this study will need to use some of this tissue, there is a small risk that it could be used up.

#### **Risks of Blood Draws**

The risks of taking blood include pain (or discomfort), possible bruising, redness or swelling at or around the point where the blood is taken, possible feeling of lightheadedness, and rare risks of fainting or infection at the point where the blood is taken.

#### **Side Effect Risks**

The drugs (and possible radiation therapy) used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drugs (and possible radiation therapy).

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

This study is looking at three chemotherapy drugs used to treat this type of cancer plus one of two study drugs. Using these drugs together may increase your side effects or may cause new side effects.

## **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Call or see your healthcare provider right away if you develop any problems listed below or the symptoms get worse.

#### For both Group 1 and Group 2:

## Possible Side Effects of Dacarbazine, Doxorubicin, Vinblastine

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Dacarbazine, Doxorubicin, Vinblastine, more than 20 and up to 100 may have:

- High blood pressure which may cause headaches, dizziness, blurred vision
- Low blood pressure which may cause feeling faint
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Nausea, vomiting, loss of appetite
- Mouth sores
- Headache
- Pain
- Muscle weakness, tiredness
- Flu-like symptoms including fever, chills, body aches, muscle pain
- Red colored urine, saliva, or sweat
- Hair loss

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Dacarbazine, Doxorubicin, Vinblastine, from 4 to 20 may have:

- Heart failure or heart attack which may cause shortness of breath, swelling of ankles, cough or tiredness which may occur years after the dose
- Abnormal heartbeat
- Stroke, which may cause paralysis, weakness
- Bleeding in the brain which may cause confusion
- Seizure
- Damage to the lungs which may cause shortness of breath
- Cancer of the bone marrow (leukemia) caused by chemotherapy
- Blood clot
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require transfusion
- Damage to the liver which may cause belly pain, bleeding, yellowing of eyes and skin
- Kidney damage which may require dialysis
- Sores in the mouth or throat
- Belly pain
- Nausea, diarrhea, vomiting, loss of appetite, constipation
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Abnormal menstrual period
- Confusion
- Numbness and tingling in fingers and toes
- Damage to the skin which may cause pain
- Swelling and redness at the site of the medication injection or area of previous radiation
- Loss of nails
- Darkening of the nail beds or skin or hands and feet

#### RARE, AND SERIOUS

In 100 people receiving Dacarbazine, Doxorubicin, Vinblastine, 3 or fewer may have:

- Severe blood infection
- Damage to hearing which may be permanent
- Increased risk of sunburn

## For Group 1 only:

#### Possible Side Effects of Nivolumab.

## **Special precautions:**

Side effects of nivolumab may happen anytime during treatment or even after your treatment has ended. Call or see your healthcare provider right away if you develop any problems listed below or the symptoms get worse.

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving nivolumab, more than 20 and up to 100 may have:

#### Tiredness

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving nivolumab, from 4 to 20 may have:

- Anemia which may require blood transfusion
- Swelling and redness of the eye
- Pain
- Diarrhea, nausea
- Dry mouth
- Fever
- Swelling and redness at the site of the medication injection
- Bruising, bleeding
- Pain or swelling of the joints
- Loss of appetite
- Reaction during or following a drug infusion which may cause fever, chills, rash

Nivolumab may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine. Signs and symptoms of colitis may include: diarrhea or increase in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly pain or tenderness.
- Skin: itching; rash, blisters including inside the mouth; loss of skin pigment
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly.
- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior decreased sex drive; weight loss or weight gain; excessive thirst or urination; dizziness or fainting.

#### RARE, AND SERIOUS

In 100 people receiving nivolumab, 3 or fewer may have:

- Swelling of arms and legs which may cause a feeling of heaviness and tightness
- Dry eyes
- Sores in the mouth which may cause difficulty swallowing
- A syndrome starting with flu-like symptoms and followed by swelling, tenderness which may cause flu-like symptoms, blurred vision, ringing in the ears, changes in hair or hair loss
- Swelling of the bowels

Nivolumab may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Visual disturbances which may cause double vision, blurred vision, or loss of vision with a chance of blindness
- A condition with high blood sugar which leads to tiredness, frequent urination, excessive thirst, headache, nausea and vomiting, and can result in coma
- Kidney problems, including nephritis and kidney failure requiring dialysis. Signs of kidney problems may include: decrease in the amount of urine, blood in your urine, ankle swelling.
- Heart problems including swelling and heart failure. Symptoms and signs of heart problem may include: Shortness of breath, swelling of the ankle and body.
- Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine
- Swelling of the brain (meningitis/encephalitis), which may cause: headache, stiff neck, confusion, sleepiness, seizures or injury to the brain which may cause headache, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs and facial muscle movement.
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Complications associated with stem cell transplant using donor stem cells (allogeneic stem cell transplant). These complications are caused by attack of donor cells on the host organs (inducing liver, skin and gut damage), and can lead to death. If you are considering an allogeneic stem transplant after participating in this study, please tell your doctor that you have received nivolumab therapy, since the risk and severity of transplant-associated complications may be increased.

#### For Group 2 only:

#### Possible Side Effects of Brentuximab vedotin

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving SGN-35 (brentuximab vedotin), more than 20 and up to 100 may have:

- Diarrhea, nausea
- Tiredness
- Numbness, tingling or pain of the arms and legs

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving SGN-35 (brentuximab vedotin), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Pain
- Constipation, vomiting
- Chills, fever
- Swelling of arms and legs
- Liver damage which may cause yellowing of the eyes and skin
- Infection, especially when white blood cell count is low
- Cold symptoms such as stuffy nose, sneezing, sore throat
- Bruising, bleeding
- Weight loss, loss of appetite
- Dizziness, headache
- Feeling of "pins and needles" in arms and legs
- Muscle weakness
- Worry
- Difficulty sleeping
- Cough, shortness of breath
- Hair loss, itching, rash
- Increased sweating

## RARE, AND SERIOUS

In 100 people receiving SGN-35 (brentuximab vedotin), 3 or fewer may have:

- Damage to the pancreas which may cause belly pain and hospitalization
- Swelling of the bowels
- Bleeding from multiple sites
- Internal bleeding which may cause black tarry stool, blood in vomit
- Blockage of internal organs which may cause difficulty swallowing, inability to pass stool
- A tear or hole in internal organs that may require surgery
- Sores in the throat
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Kidney damage which may require dialysis
- Damage to the lungs which may cause shortness of breath
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

For men: Many cancer treatments damage the cells that grow into sperm. Sometimes these cells recover, but sometimes they do not. We don't know for certain how your treatment will affect your future fertility. You may not be thinking about being a father right now. However, one day this may be important to you. Sperm banking is the collection, freezing, and storage of sperm for possible use in the future. Sperm banking before treatment may increase your chance of having a biological child in the future using your own sperm.

**Possible Side Effects of Pegfilgrastim** 

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving Pegfilgrastim, more than 20 and up to 100 may have:

• Pain in bone

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Pegfilgrastim, from 4 to 20 may have:

- Anemia which may cause tiredness, or may require transfusion
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Damage to the lungs which may cause shortness of breath

#### RARE, AND SERIOUS

In 100 people receiving Pegfilgrastim, 3 or fewer may have:

• Rupture of the spleen causing sudden or severe pain in the left side of abdomen spreading up to your shoulder

**Possible Side Effects of Filgrastim** 

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Filgrastim, more than 20 and up to 100 may have:

- Nose bleed
- Anemia which may require transfusion
- Pain
- Diarrhea
- Fever
- Tiredness
- Hair loss

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Filgrastim, from 4 to 20 may have:

- Fluid in the organs which may cause low blood pressure, shortness of breath, swelling of ankles
- Damage to the lungs which may cause shortness of breath
- Internal bleeding which may cause coughing up blood
- Cough
- Swelling or tenderness of vessels
- Headache

## RARE, AND SERIOUS

In 100 people receiving Filgrastim, 3 or fewer may have:

• Rupture of the spleen causing sudden or severe pain in the left side of abdomen spreading up to your shoulder

The study drugs could interact with other drugs. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

## **Possible Side Effects of Radiation Therapy**

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving radiation therapy, 20 to 100 may have:

- Reddening, tanning, or peeling of the skin
- Mild pain
- Hair loss
- Tiredness
- Diarrhea, nausea
- Anemia, which may require transfusion
- Infection, especially when white blood cell count is low

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving radiation therapy, 4 to 20 may have:

- Thickening and numbness of the skin
- Sores or ulcers on the skin or near the cancer location
- Permanent hair loss
- Bleeding from the skin
- Sores in mouth which may cause difficulty swallowing

## RARE, AND SERIOUS

In 100 people receiving radiation therapy, 3 or fewer may have:

- Damage to internal organs
- Abnormal opening in internal organs which may cause pain and bleeding

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

## What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications (prescribed by your doctor or purchased over-the-counter) and supplements (such as vitamins or herbs) you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.

**For women:** Do not get pregnant or breastfeed while taking part in this study or for 6 months after you receive the last dose of study drug or after you receive the last dose of radiation therapy (if applicable).

For men: Do not father a baby while taking part in this study or for 7 months after your last dose of study drug or for 6 months after your last dose of radiation therapy (if applicable). If you will be receiving brentuximab vedotin (Group 2), ask your doctor about sperm banking.

**For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 7 months after your last dose of study drug.

# What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer.

This includes:

- the costs of tests (including blood tests, such as thyroid function testing), exams, procedures, and drugs that you get during the study to monitor your safety and prevent and treat side effects.
- the costs of getting the study drugs nivolumab (Group 1), brentuximab vedotin (Group 2), doxorubicin (Group 1 and 2), vinblastine (Groups 1 and 2), dacarbazine (Groups 1 and 2) and filgrastim or pegfilgrastim (for all patients in Group 2 and for patients in Group 1, if recommended by your doctor) ready and giving it to you.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You or your insurance provider will not have to pay for the nivolumab while you take part in this study.

You or your insurance provider will be responsible for all other costs, including the cost of the blood tests (including thyroid function testing), the costs of imaging (including PET-CT scans), the cost of the drugs (including brentuximab vedotin, doxorubicin, vinblastine, dacarbazine, and pegfilgrastim or filgrastim), and the costs of getting the study drugs (including nivolumab) ready to give to you.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat the cancer. You may:

- Have more travel costs.
- Need to take more time off work or school.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor (SWOG Cancer Research Network) and any company supporting the study drug now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA, Health Canada and the groups these agencies work with to review research.
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

## Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| | • |
|---|---|
| You can talk to the study doctor aboreport side effects or injuries. Conta | the study doctor (insert name of |
| study doctor[s]) atappropriate). | (insert telephone number and email address if |
| For questions about your rights w | hile in this study, call the |
| (insert name of organization or cen | er) Institutional Review Board at |
| (insert telephone number). (Note to | Local Investigator: Contact information for patient |
| representatives or other individuals | at a local institution who are not on the IRB or research |
| team but take calls regarding clinic | al trial questions can also be listed here.) |

# Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with cancer in the future.

The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say 'no' to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

# Optional Sample Collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

## **Unknown future studies**

If you choose to take part in this optional study, a sample of tissue from your biopsy at time of cancer diagnosis will be stored and samples of your blood will be collected and stored. Storing samples for future studies is called "biobanking". The Biobank is being run by Nationwide Children's Hospital and supported by the National Cancer Institute. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your blood and tissue samples.

This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes.

If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

## What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. About 4 teaspoons of blood will be collected from a vein in your arm at 3-4 timepoints: Cycle 1/Day 1, Cycle 3/Day 1, at time of completion of treatment (after Cycle 6 or when you stop receiving study drug), and at the time the Hodgkin Lymphoma gets worse (if that happens).
- 2. A sample from the tissue that was collected at the time of the cancer diagnosis will be sent to the biobank. If your cancer gets worse (progresses), then a sample of the tissue that is taken at the time of progression (as part of the usual care for cancer) will also be sent to the biobank.
- 3. Your sample will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 4. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 5. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

## What are the risks in this optional sample collection?

- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/

If you choose to take part in the **Optional Image Collection for Storage for Possible Future Studies**, then the PET-CT scans which were collected as part of the usual care for your cancer at 3 timepoints (prior to beginning the study, after completion of Cycle 2, and 4-8 weeks after Cycle 6, Day 15) will be stored for future unknown research studies. You will not receive any extra scans for research purposes alone. The future research review of your scans will only be used for research and will not to guide your medical care.

## What are the risks in this optional image collection?

- Your privacy is very important to the study researchers. They will make every effort to protect it.
- There is a risk that someone outside of the research study could get access to your study records or trace information in a database back to you. They could use that information in a way that could harm you. Researchers believe the chance that someone could access and misuse your information is very small. However, the risk may increase in the future as people find new ways of tracing information.

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

What are the benefits to taking part in this optional sample or image collection?

You will not benefit from taking part.

The researchers, using the samples or images from you and others, might make discoveries that could help people in the future.

# Are there any costs or payments to this optional sample or image collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

| What if I change my mind about this optional sample collection? |
|---|
| If you decide you no longer want your samples to be used, you can call the study doctor |
| (insert name of study doctor for main trial) at |
| (insert telephone number and email address of study doctor for main) who will let the biobank know. Then, any sample that remains in the biobank will be <i>trial</i> destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers. |
| What if I change my mind about this optional image collection? |
| If you decide you no longer want your images to be used, you can call the study doctor |
| (insert name of study doctor for main trial) at |
| (insert telephone number and email address of study doctor for main trial) who will let the image bank know. Then, your scans will be destroyed and will no longer be used in any future |
| research. If your images (scans) or related health information were previously shared with |
| researchers, then the scans will be retained by those researchers for the duration required by the research protocol, and your scans/images will still be used in the research outcomes. |
| What if I have questions about this optional sample or image collection? |
| If you have questions about the use of your samples for research, contact the study doctor |
| (insert name of study doctor for main trial) at |
| (insert telephone number and email address of study doctor for main trial). |

Please circle your answer below to show if you would or would not like to take part in each optional study:

# Samples for unknown Future Research Studies

My samples and related information may be kept in a Biobank for use in future health research.

YES NO

# Images (PET-CT scans) for unknown Future Research Studies

My images and related information may be stored for use in future health research.
YES NO

## **Contact for Future Research**

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

This is the end of the section about optional studies.

# My Signature Agreeing to Take Part in the Study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the main study and any additional studies where I circled 'yes'. I also agree to take part in any additional studies where I circled "yes".

| Participant's signature (or legally authorized representative) | |
|---|---|
| Date of signature | |
| For non-COG sites, Signature of person(s) conducting the inf | ormed consent discussion |
| Date of signature | |
| Parent/Guardian signature | _ |
| Date of signature | |
| Parent/Guardian signature | _ |
| Date of signature | |
| For COG patient registration, Physician/PNP obtaining conso | ent |
| Date of signature | |